CLINICAL TRIAL: NCT03153189
Title: Correlates of Physical Activity With Anthropometric Traits, Mental Health and Quality of Life in College Women of Manipal University
Brief Title: Correlates of Physical Activity With Quality of Life in College Women of Manipal University
Acronym: PA
Status: Completed | Type: Observational
Sponsor: Manipal University (Other)
Responsible Party: Principal Investigator, Hiral Chauhan, Postgraduate, Manipal University
Other Study IDs: REF/2017/05/014211
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Physical Activity
Keywords: PA,menatal health,QOL
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To find out the relationship between physical activity and

* self-esteem,
* sleep quality,
* anxiety & depression,
* body fat percentage,
* quality of life, in college females

DETAILED DESCRIPTION:
* After receiving approval from the Institutional Research Committee and Institutional Ethical Committee clearance.
* Advertisement of the research project will be done via the Head of Department of each faculty of the university
* Subjects will be recruited on a voluntary basis and a written informed consent will be obtained after the research idea is explained.
* Demographics of each participant will be obtained
* Each of the following questionnaires will be administered:

Depression, Anxiety and Stress Scale (DASS-21) Rosenberg Self-Esteem Scale Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) Pittsburgh Sleep Quality Index (PSQI) International Physical Activity Questionnaire-Long Form (IPAQ)

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* age group 18-25
* Indian ethnicity

Exclusion Criteria:

* Known cardio-respiratory symptoms and musculoskeletal disorders curtailing form physical activity in the last 3 months, known thyroid dysfunction, known anxiety-depression disorders, recent surgery (last 3months), polycystic ovary disease (PCOD), polycystic ovary syndrome (PCOS) & pregnancy.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female who all under 18 -25 yr old and are a student of Manipal University.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire-Long Form (IPAQ) | immediate
  score of the questionnaire in MET/hr

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sport Science Medicine and Research, Udupi, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anjana RM, Pradeepa R, Das AK, Deepa M, Bhansali A, Joshi SR, Joshi PP, Dhandhania VK, Rao PV, Sudha V, Subashini R, Unnikrishnan R, Madhu SV, Kaur T, Mohan V, Shukla DK; ICMR- INDIAB Collaborative Study Group. Physical activity and inactivity patterns in India - results from the ICMR-INDIAB study (Phase-1) [ICMR-INDIAB-5]. Int J Behav Nutr Phys Act. 2014 Feb 26;11(1):26. doi: 10.1186/1479-5868-11-26. PMID 24571915
- [Result] Rimer J, Dwan K, Lawlor DA, Greig CA, McMurdo M, Morley W, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD004366. doi: 10.1002/14651858.CD004366.pub5. PMID 22786489
- [Result] Backhaus J, Junghanns K, Broocks A, Riemann D, Hohagen F. Test-retest reliability and validity of the Pittsburgh Sleep Quality Index in primary insomnia. J Psychosom Res. 2002 Sep;53(3):737-40. doi: 10.1016/s0022-3999(02)00330-6. PMID 12217446